CLINICAL TRIAL: NCT00284284
Title: Investigation of the Added Value of a Big Toe Hinged Brace for the Treatment of Hallux Rigidus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/171
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Hallux Rigidus
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Use of a rehabilitation brace

SUMMARY:
Comparison of the added value of a rehabilitation brace to standard rehabilitation by physiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Hallux rigidus

Exclusion Criteria:

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Mobility of the big toe joint

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be